CLINICAL TRIAL: NCT04472169
Title: Value of Emicizumab Monitoring With UPLC-MS/MS for Bleeding Risk Prediction in Severe Hemophilia A
Brief Title: UPLC-MS/MS Monitoring of Emicizumab Therapy
Acronym: EMICARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_75; 2020-A00584-35 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Hemophilia A
Keywords: Drug monitoring; Severe Hemophilia A; Emicizumab
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, poor-platelet plasma, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe haemophila A patients with or without inhibitors

SUMMARY:
Emicizumab is a monoclonal bispecific antibody with a terminal half-life of 28 days which is now licensed in the treatment of severe haemophilia A with or without inhibitors. Some heterogeneity in residual emicizumab concentrations have been reported according to age, body mass index or drug therapeutic regimen. Some cases of neutralizing antidrug antibodies have been also reported. Whether monitoring emicizumab plasma concentration could predict the residual bleeding risk under emicizumab is unknown. As conventional coagulation assays are not adapted for emicizumab monitoring, this study aims to assess the value of monitoring residual emicizumab plasma concentration by UPLC-MS/MS in bleeding risk prediction.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child with Clinical diagnosis of severe hemophilia A (FVIII activity < 1%) with or without inhibitor
* Clinical indication to emicizumab therapy

Exclusion Criteria:

* Refusal to give informed consent
* acquired hemophilia A
* other inherited or acquired bleeding disorder
* bodyweight < 10 kgs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients with severe hemophilia A will be included in the study on 2 french Hemophilia Treatement Centers (CHU Lille and CHU Caen)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Area under the curve ROC of Residual plasma level of emicizumab | At Week 5 (end of emicizumab loading period)
  At least one clinically significant bleeding (defined as any bleeding treated with FVIII, rFVIIa or aPCC) from loading period completion (week 5) to the end of study, an average of 1 year

SECONDARY OUTCOMES:
Residual plasma level of emicizumab measured by UPLC-MS/MS | At Week 5 (end of emicizumab loading period)
  At least one hemarthrosis from loading period completion (week 5) to the end of study, an average of 1 year
Residual plasma level of emicizumab measured by UPLC-MS/MS | At each breakthrough bleeding until end of study
  Post-traumatic or spontaneous nature of bleeding event
Residual plasma level of emicizumab (UPLC-MS/MS dosing) | At Week 5 and at each breakthrough bleeding until end of study
  Emicizumab FVIII-like activity (chromogenic FVIII BIOPHEN™assay system with emicizumab calibration)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Rauch, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - CHU de Caen, Caen
  - Institut Coeur-Poumon, Pôle d'Hématologie-Transfusion, CHU, Lille